CLINICAL TRIAL: NCT06647524
Title: Pilot fMRI Studies of Aging-Related Effects of THC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Biopharmaceutical Research Company (Unknown); Bloom Labs Cannabis Solutions (Unknown)
Responsible Party: Principal Investigator, Godfrey Pearlson, Professor of Psychiatry and of Neuroscience, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2000032428; HHC-2024-0186 (Other: Hartford Healthcare)
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: THC
Keywords: Memory Impairment; Learning Impairment
MeSH Terms: conditions — Memory Disorders | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The dose will be portioned by the unblinded co-investigator to assure each participant receives the correct dose.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- THC then Placebo (Experimental): Participants in this arm will receive THC then placebo in a 2-session per subject double-blind, random assignment, placebo-controlled counterbalanced design. (Participants randomized to receive THC in the first session will receive placebo at the 2nd session.) Sessions will be scheduled at least one week apart. Tasks tapping each of the major cognitive memory-related domains will be performed in the MRI scanner, to reveal the relevant underlying circuitry and its disruption by drug using functional MRI.
  Interventions: Drug: THC; Drug: Placebo
- Placebo then THC (Placebo Comparator): Participants in this arm will receive placebo then THC in a 2-session per subject double-blind, random assignment, placebo-controlled counterbalanced design. (Participants randomized to receive placebo in the first session will receive THC at the 2nd session.) Sessions will be scheduled at least one week apart. Tasks tapping each of the major cognitive memory-related domains will be performed in the MRI scanner, to reveal the relevant underlying circuitry and its disruption by drug using functional MRI.
  Interventions: Drug: THC; Drug: Placebo

INTERVENTIONS:
Drug: THC — Participants will be administered 0.5g of vaporized THC cannabis (12% THC cannabis)
Drug: Placebo — Participants will be administered identical plant material from which all THC has been removed by solvent extraction.

SUMMARY:
The purpose of this study is to begin investigating acute impairment of various forms of memory and learning by Tetrahydrocannabinol (THC) in cannabis (CNB) compared to placebo, in a 2-session per subject double-blind, random assignment, placebo-controlled counterbalanced design in young to middle-aged adults.

DETAILED DESCRIPTION:
Tasks tapping each of the major cognitive memory-related domains will be performed in the MRI scanner, to reveal the relevant underlying circuitry and its disruption by drug using functional MRI.

On an initial Screening Visit, regular or novice cannabis (CNB) users will undergo informed consent, clinical assessment (to fully evaluate inclusion/exclusion criteria), cognitive/personality assessment, and a structural MRI scan.

At each assessment, subjects will provide subjectively-rated CNB intoxication using a verbal analog scale, complete 2 fMRI paradigms within ~1.5 hours: a) Card Guessing task and b) Complex Working Memory Span, and complete the computer-based Effort Expenditure for Reward Task within ~2 hours. These tests will be counterbalanced across subjects and sessions to minimize order and fatigue effects. Breaks will be standardized in a private environment and snacks/meals provided. Bathroom visits given as needed. Subjects will be supervised at all times by study staff and vital signs monitored. On assessment days, participants will remain at the Olin NRC until they report no subjective intoxication, and are observed by study staff to be no longer objectively intoxicated, then use taxi or Uber transportation home.

ELIGIBILITY:
Inclusion Criteria:

* CNB use within past 2 years and felt "high" when used.
* Able to read, speak, and understand English.
* Able and willing to provide written informed consent, and willing to commit to the study protocol.

Exclusion Criteria:

* Current marijuana tolerance, desire to cut down, or cravings to use during periods of abstinence.
* Positive screen for drug or alcohol (except CNB) on test day will result in rescheduling the appointment
* History of adverse effects with CNB
* CNB users who are abstaining
* IQ <80 on the Wechsler Abbreviated Scale of Intelligence
* Inability to comprehend written instructions using the WRAT 4 reading achievement test
* Pregnant, breastfeeding, and ineffective birth control methods
* Unable or unsafe to have an MRI
* Serious medical, neuro-ophthalmological, or neurological illness (e.g. cancer, seizure disorders, encephalopathy
* History of head trauma with loss of consciousness > 30 minutes or concussion lasting 30 days
* Focal brain lesion seen on structural MRI
* Any medical/neurological condition that could compromise neurocognitive performance (e.g. epilepsy, multiple sclerosis, fetal alcohol syndrome)
* Anyone deemed unsafe to study personnel for any reason
* Hearing loss such that subject cannot hear sounds at the levels (dB) or pitches (Hz) to be used in the study
* Significant pain and/or reduced mobility in the arms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The Complex Working Memory Span (CWMS) Task- Items Recalled | At sessions 1 and 2 while under fMRI, immediately post drug administration
  CWMS Task assesses immediate plus delayed recall and working memory by assessing working memory capacity by presenting a list of stimuli to be recalled while simultaneously performing a secondary task. This task uses a fully crossed design which includes both same-domain CWMS conditions (e.g. verbal storage combined with verbal processing) as well as cross-domain CWMS conditions (e.g., verbal storage combined with spatial processing). Mean number of total items recalled.
The Complex Working Memory Span (CWMS) Task- fMRI measure | At sessions 1 and 2 while under fMRI, immediately post drug administration
  CWMS Task assesses immediate plus delayed recall and working memory by assessing working memory capacity by presenting a list of stimuli to be recalled while simultaneously performing a secondary task. This task uses a fully crossed design which includes both same-domain CWMS conditions (e.g. verbal storage combined with verbal processing) as well as cross-domain CWMS conditions (e.g., verbal storage combined with spatial processing). BOLD signal Infrontal lobe.
The Effort Expenditure for Reward Task (EEfRT) | At sessions 1 and 2 immediately post drug administration
  (EEfRT) is an out-of-scanner measure of effort-based decision-making that utilizes a choice model ("easy-task" or "hard-task") in response to varying monetary rewards. This task assesses motivation in relation to reward magnitude, implicating the activation or suppression of dopaminergic pathways in the nucleus accumbens (NAcc). Percentage of hard-task choices across all levels of probability is calculated from all hard choices. Lower percentages of hard task choices indicate decreased motivation.
The Card-Guessing fMRI task | At sessions 1 and 2 while under fMRI, immediately post drug administration
  The Card-Guessing fMRI task (28) will be used to investigate the effects of acute THC intoxication on decision-making, risk-taking, and reward processing. This task involves various trial types including win, loss, disappointment, and relief, to assess how THC affects reward expectancy and prediction error processing during decision-making presented as the fMRI blood-oxygen-level-dependent (BOLD) signal in response to card-guessing task.
The Zibrio SmartScale | At sessions 1 and 2 while under fMRI, immediately post drug administration
  The Zibrio SmartScale aggregates balance data to create a "Balance Score", which assesses postural sway with respect to balance ability and fall risk. Total score range 1 and 10. A lower score indicates a higher risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Pearlson, M.D, Principal Investigator — Founding Director, Olin Neuropsychiatry Center; Yale University
Locations (1):
- Olin Neuropsychiatric Research Center at Hartford Healthcare, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No